CLINICAL TRIAL: NCT02126319
Title: Facilitating Participation in a Prostate Cancer Family Risk Assessment Program
Brief Title: Facilitating Participation in a Prostate Cancer Risk Assessment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB97-811; TPRB-98-266-01-PBP (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2014-03-24; First posted 2014-04-30 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
Keywords: Cognitive-affective preparation; prostate cancer counseling
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Affective Preparation (Experimental): Forty five minute cognitive-affective preparation session, wherein individuals were encouraged to experience and self-assess their personal reactions to the information they had just received about their prostate cancer risk status, and to anticipate ("pre-live") and role play their potential psychological reactions to normal and abnormal test results and associated follow-up diagnostic and management recommendations. Combined with standard Prostate Risk Assessment Program (Group Prostate Cancer Education Session, Individual Counseling, Screening feedback)
  Interventions: Behavioral: Cognitive Affective preparation
- General Health Education (Active Comparator): A general health educational comparison session administered by research staff in order to equate for factual content, time, and attention. Participants in this session received information of relevance to men at risk for Pca, focusing on recommendations for general health (i.e., diet, exercise, alcohol use, and smoking) and were encouraged to freely probe, explore, and discuss their own attitudes, beliefs, expectations, and feelings about these topics in an interactive format. Combined with standard Prostate Risk Assessment Program (Group Prostate Cancer Education Session, Individual Counseling, Screening feedback)
  Interventions: Behavioral: General Health Education

INTERVENTIONS:
Behavioral: Cognitive Affective preparation — Forty five minute cognitive-affective preparation session, wherein individuals were encouraged to experience and self-assess their personal reactions to the information they had just received about their prostate cancer risk status, and to anticipate ("pre-live") and role play their potential psychological reactions to normal and abnormal test results and associated follow-up diagnostic and management recommendations. Combined with standard Prostate Risk Assessment Program (Group Prostate Cancer Education Session, Individual Counseling, Screening feedback)
  Arms: Cognitive Affective Preparation
Behavioral: General Health Education — A general health educational comparison session administered by research staff in order to equate for factual content, time, and attention. Participants in this session received information of relevance to men at risk for Pca, focusing on recommendations for general health (i.e., diet, exercise, alcohol use, and smoking) and were encouraged to freely probe, explore, and discuss their own attitudes, beliefs, expectations, and feelings about these topics in an interactive format. Combined with standard Prostate Risk Assessment Program (Group Prostate Cancer Education Session, Individual Counseling, Screening feedback)
  Arms: General Health Education

SUMMARY:
The purpose of this study was to examine whether a cognitive-affective preparation was more beneficial, in general, and more specifically for certain subgroups, such as African-American men and individuals with high monitoring style.

DETAILED DESCRIPTION:
High risk men enrolling in a state of the science Prostate Cancer Risk Assessment Program (N = 128) underwent a Pca counseling visit immediately followed by either a cognitive-affective preparation (CAP) session designed to help men process the information they received or a general health education session to control for time and attention (comparison group). All men chose to participate in Pca screening.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men, 34 and 69 years of age, at least one first or second degree relative with prostate cancer

OR

* African American men, 35 and 69 years of age

Exclusion Criteria:

* cancer diagnosis
* difficulty communicating in English
* impaired competency to give informed consent.

Ages: 34 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 1998-10; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Miller, Ph.D., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Affective Preparation | General Health Education
Started | 61 | 67
Completed | 40 | 43
Not Completed | 21 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Affective Preparation | General Health Education | Total
Number analyzed (Participants) | 61 | 67 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.21 (8.86) | 47.61 (8.81) | 47.42 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 67 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 33 | 66
  White | 28 | 34 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
family history of Pca [Number; unit: participants] — Baseline information regarding family history for prostate cancer was incomplete. A man was considered as having a positive family history for prostate cancer if Data at baseline was incomplete regarding this variable (20 men for the General Health Education Group and 16 men for the Cognitive Affective Preparation Group).
  participants
    With positive family history | 47 | 58 | 105
    No family history | 14 | 9 | 23
Pca related knowledge [Mean (Standard Deviation); unit: units on a scale] — Knowledge about Pca risk was measured using an eight item scale prepared for this study. It consisted of true/false items (e.g., "An abnormal DRE and/or PSA could be the result of conditions other than prostate cancer"). Correct responses received a value of one, whereas false responses received a zero. Values ranged between zero and eight, with higher values indicating higher knwoledge.
  units on a scale | 6.53 (1.40) | 6.23 (1.39) | 6.37 (1.40)
Pca related perceived risk [Mean (Standard Deviation); unit: units on a scale] — Perceived risk of Pca was assessed using four items where participants were asked to estimate their prostate cancer risk in general (e.g., "Do you feel as though you are the kind of person who is likely to develop prostate cancer?") or comparing themselves to other men at risk for Pca (e.g., "Given your ethnicity, what are your chance of getting prostate cancer?") on a five-point scale (Lerman et al., 1996). Reported means are based on a scale from one to five. Higher scores indicate higher Pca perceived risk i.e. 1=much lower risk; 5=much higher risk. Cronbach's alpha for the scale was 0.83.
  units on a scale | 3.10 (0.87) | 3.25 (0.77) | 3.18 (0.82)
Pca related positive expectancies [Mean (Standard Deviation); unit: units on a scale] — Positive expectancies regarding the effects of screening were assessed using two items on a five-point scale ("Regular screening will ensure that I stay healthy" and "Regular screening will prolong my life"). Questionnaire items were author-constructed, based on prior work and cognitive-affective theory (Miller et al., 1996). Reported means are based on a scale from one to five. Higher scores indicate more Pca related positive expectancies. Cronbach's alpha for the scale was 0.76.
  units on a scale | 3.86 (1.09) | 3.97 (0.91) | 3.92 (0.99)
Pca related negative expectancies [Mean (Standard Deviation); unit: units on a scale] — Negative expectancies related to Pca screening comprised five items and assessed the costs and risks of screening, in terms of time and effort, fears of discrimination, insurance and employment, and financial concerns on a five-point scale (e.g., "Screening may have a negative impact on my health insurance"). Questionnaire items were author-constructed, based on prior work and cognitive-affective theory (Miller et al., 1996). Reported means are based on a scale from one to five. Higher scores indicate more negative expectancies. Cronbach's alpha for the scale was 0.80.
  units on a scale | 1.72 (0.78) | 1.72 (0.78) | 1.72 (0.78)
Pca related intrusive ideation [Mean (Standard Deviation); unit: units on a scale] — Intrusive ideation related to prostate cancer risk was assessed using the Impact of Events Scale (IES) (Horowitz et al., 1979). This instrument has been used extensively in the cancer literature (Schwartz et al., 2002). Only the intrusive ideation subscale was used in this study. The range of possible values is 0 to 35. Higher scores indicate higher level of intrusive ideation. Cronbach's alpha for the intrusion subscale in the present study was 0.82. Because of high skewness, a median split was used to create a high and a low group.
  units on a scale | 4.51 (5.81) | 3.33 (4.32) | 3.89 (5.10)
Monitoring attentional style [Number; unit: participants] — Monitoring attentional style was assessed at baseline using the Monitoring Style Subscale (MBSS; Miller, 1987), which measures attentional responses to four structured stress-evoking scenarios. Each scenario is followed by four possible monitoring responses. Participants endorse all the responses that apply to them. A total monitoring score (range 0-16) is computed for each participant by summing the number of monitoring responses endorsed within each of the four scenarios. A median split was used to create a high (greater than 9) and a low (less or equal to 9) monitoring group.
  participants
    High | 28 | 31 | 59
    Low | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Pca Risk-related Knowledge
Description: Knowledge about Pca risk was measured using an eight item scale prepared for this study. It consisted of true/false items [e.g., "An abnormal digital rectal examination (DRE) and/or prostate-specific antigen (PSA) could be the result of conditions other than prostate cancer"]. Correct responses received a value of one, whereas false responses received a zero. Values ranged between zero and eight. Higher score means better knowledge of risk and issues.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 38 | 42
units on a scale | 6.92 (1.02) | 7.19 (0.99)

2. Primary Outcome: Pca Perceived Risk
Description: Perceived risk of Pca was assessed using four items where participants were asked to estimate their prostate cancer risk in general (e.g., "Do you feel as though you are the kind of person who is likely to develop prostate cancer?") or comparing themselves to other men at risk for Pca (e.g., "Given your ethnicity, what are your chance of getting prostate cancer?") on a five-point scale (Lerman et al., 1996). Reported means are based on a scale from one to five (based on the average of the four items). Cronbach's alpha for the scale was 0.83. A higher score indicates higher Pca perceived risk.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 42 | 46
units on a scale | 3.23 (0.82) | 2.98 (0.82)

3. Primary Outcome: Pca-related Positive Expectations
Description: Positive expectations regarding the effects of screening were assessed using two items on a five-point scale ("Regular screening will ensure that I stay healthy" and "Regular screening will prolong my life"). Questionnaire items were author-constructed, based on our prior work and cognitive-affective theory (Miller et al., 1996). Reported means are based on a scale from one to five (average of the two items). Cronbach's alpha for the scale was 0.76. Higher score indicates more positive expectations.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 42 | 49
units on a scale | 3.66 (1.16) | 4.07 (0.79)

4. Primary Outcome: Negative Expectations Regarding Pca Risk
Description: Negative expectations related to Pca screening comprised five items and assessed the costs and risks of screening, in terms of time and effort, fears of discrimination, insurance and employment, and financial concerns on a five-point scale (e.g., "Screening may have a negative impact on my health insurance"). Questionnaire items were author-constructed, based on our prior work and cognitive-affective theory (Miller et al., 1996). Reported means are based on a scale from one to five (average of five items). Cronbach's alpha for the scale was 0.80. A higher score indicates more negative expectations.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 41 | 49
units on a scale | 1.47 (0.57) | 1.53 (0.70)

5. Primary Outcome: Pca Related Intrusive Ideation
Description: Intrusive ideation related to prostate cancer risk was assessed using the Impact of Events Scale (IES) (Horowitz et al., 1979). The full scale consists of two subscales, intrusive ideation and avoidant ideation. In this study only the intrusive ideation subscale was used. The instrument has been used extensively in the cancer literature (Schwartz et al., 2002). Values range from 0 to 35, with higher values indicating a higher level of intrusive ideation. Cronbach's alpha for the intrusion subscale in the present study was 0.82. Because of high skewness, a median split was used to create a high intrusive ideation group and a low intrusive ideation group.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 42 | 48
units on a scale | 3.64 (5.97) | 3.31 (5.30)

6. Primary Outcome: Pca Risk-related Knowledge
Description: as for outcome 1
Time Frame: six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 39 | 40
units on a scale | 7.03 (1.27) | 7.03 (1.19)

7. Primary Outcome: Pca Perceived Risk
Description: as for outcome 2
Time Frame: six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 39 | 40
units on a scale | 2.99 (.82) | 3.13 (.83)

8. Primary Outcome: Pca-related Positive Expectations
Description: as for outcome 3
Time Frame: six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 40 | 45
units on a scale | 3.85 (1.10) | 3.70 (0.88)

9. Primary Outcome: Negative Expectations Regarding Pca Risk
Description: Negative expectations related to Pca risk screening comprised five items and assessed the costs and risks of screening, in terms of time and effort, fears of discrimination, insurance and employment, and financial concerns on a five-point scale (e.g., "Screening may have a negative impact on my health insurance"). Questionnaire items were author-constructed, based on our prior work and cognitive-affective theory (Miller et al., 1996). Reported means are based on a scale from one to five (average of five items). Cronbach's alpha for the scale was 0.80. A higher score indicates more negative expectations.
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 39 | 44
units on a scale | 2.12 (.58) | 2.08 (0.54)

10. Primary Outcome: Pca Related Intrusive Ideation
Description: Intrusive ideation related to prostate cancer risk was assessed using the Impact of Events Scale (IES) (Horowitz et al., 1979). The full scale consists of two subscales, intrusive ideation and avoidant ideation but only the intrusive ideation subscale was used in the present study. The instrument has been used extensively in the cancer literature (Schwartz et al., 2002). Cronbach's alpha for the intrusion subscale in the present study was 0.82. Values range from zero to 35, with higher values indicating higher level of intrusive ideation. Because of high skewness, a median split was used to create a high intrusive ideation group and a low intrusive ideation group.
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Affective Preparation | General Health Education
Number analyzed (Participants) | 39 | 45
units on a scale | 3.85 (4.92) | 2.62 (4.89)

ADVERSE EVENTS:
Time Frame: Between October 1998 and April 2002. Six months follow-up.
Arm/Group | Cognitive Affective Preparation | General Health Education
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/67
Other Adverse Events (participants affected / at risk) | 0/61 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No